CLINICAL TRIAL: NCT01117038
Title: A Phase I, Double-Blind, Randomized, Placebo-Controlled, Two-Period, Two-Cohort Crossover Study to Assess the Potential Interaction of Avanafil on the Pharmacokinetic and/or Hemodynamic Effects of Enalapril or Amlodipine in Male Subjects
Brief Title: Drug Interaction Study of Avanafil and Enalapril or Amlodipine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Wesley Day, Vivus, Inc.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-019
Record Dates: First submitted 2010-04-23; First posted 2010-05-05 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Erectile Dysfunction
Keywords: ED; Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — avanafil; Enalapril; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- enalapril and avanafil (Experimental)
  Interventions: Drug: avanafil and enalapril
- amlodipine and avanafil (Experimental)
  Interventions: Drug: avanafil and amlodipine

INTERVENTIONS:
Drug: avanafil and enalapril — enalapril twice a day for 11 days avanafil/placebo once a day for 2 days
  Arms: enalapril and avanafil
Drug: avanafil and amlodipine — amlodipine 5mg once a day for 16 days avanafil/placebo once a day for 3 days
  Arms: amlodipine and avanafil

SUMMARY:
The purpose of this study is to determine the change in the blood pressure and pulse rate, pharmacokinetics and the safety when avanafil is taken with either enalapril or amlodipine.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily consent to participate in the study (informed consent form [ICF] must be signed and dated prior to any study related assessments).
2. Adult male subjects of 40 to 65 years of age, inclusive.
3. A body weight of at least 50 kg and a body mass index (BMI) between 18 and 32 kg/m2, inclusive [BMI will be calculated as weight in kg/(height in m)2].
4. Subjects are able to communicate with the Investigator, and to understand and comply with all requirements of study participation.
5. Medically healthy, with no clinically significant screening results (e.g., laboratory profiles, medical histories, ECGs, physical examinations, etc.), in the opinion of the Investigator.

Exclusion Criteria:

1. A history or presence of significant cardiovascular (including thromboembolic disorders), neurological, hematological, psychiatric, hepatic, gastrointestinal, pulmonary, endocrine, immunologic, or renal disease, or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs or place the subjects at increased risk as determined by the Investigator.
2. Any clinically significant laboratory abnormalities as judged by the Investigator.
3. A predisposition to priapism, such as subjects with sickle cell disease or blood dyscrasias.
4. Known history of cardiovascular or cerebrovascular event, or any history of angina.
5. History of fainting or vasovagal hypotension.
6. History or ECG evidence of any high-risk arrhythmia or ECG judged by the Investigator to be clinically significant.
7. Hypertrophic obstructive or other clinically significant cardiomyopathy, moderate or severe cardiac valvular disease.
8. Subjects whose pulse is lower than 50 bpm at screening.
9. Acute illness, especially any infection, within 2 weeks of dosing.
10. Supine systolic blood pressure </= 100 or >/= 140 mmHg; supine diastolic blood pressure </= 50 or >/= 95 mmHg at screening (2 rechecks are allowed).
11. Subjects with orthostatic hypotension (as evidenced by a reduction of 30 mmHg or more in systolic blood pressure, reduction of 20 mmHg or more in diastolic blood pressure, or evidence of cerebral hypoperfusion upon standing from a seated position).
12. Any history of bipolar disorder or psychosis, history of psychiatric hospitalization, greater than one lifetime episode of major depression.
13. Hemoglobin < 12.0 g/dL.
14. Positive urine drug test, positive urine alcohol test, or positive urine cotinine test at screening or at check-in on Day -1.
15. Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV) at screening.
16. Any history or presence of alcoholism or drug or substance abuse within 18 months or as defined by the Investigator.
17. Allergy to or previous adverse events with PDE5 inhibitors, ACE inhibitors, calcium channel blockers, or their constituents.
18. Use of any prescription or over-the-counter (OTC) medication, including herbal products, within the 14 days prior to Day 1 and throughout the study. Up to 2 g per day of acetaminophen is allowed at the discretion of the Investigator.
19. Use of any drug in Appendix 1 (drugs known to interfere with metabolism by the CYP450 3A4 enzyme) within 30 days prior to Day 1.
20. Blood donation or significant blood loss within 56 days prior to Day 1.
21. Plasma donation within 14 days prior to Day 1.
22. Any use of tobacco or nicotine products within 6 months prior to Day 1.
23. Any subject who received an investigational drug within 30 days or six half-lives, whichever is longer, prior to Day 1.
24. Involvement in the planning and conduct of the study (applies to both VIVUS or designee staff, or staff at the investigational site).
25. Previously participated in a trial with avanafil.
26. Subjects who report having difficulty swallowing tablets, capsules, etc.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To measure the change in standing blood pressure after dosing | -0.5, -0.25, -0.17, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10 and 22 hours

SECONDARY OUTCOMES:
To measure the pharmacokinetic parameters of taking avanafil with enalapril | before dosing and after dosing at the hours of 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36, 48
  AUCc-tau Cmax Cmin Tmax AUC0-t AUC0-inf t1/2 Kel
To measure the change in sitting and lying blood pressure and pulse rate after dosing | -0.5, -0.33, -0.17, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10 and 22 hours
To determine the effects of enalapril on blood pressure and pulse rate | -0.5, -0.33, -0.17, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10 and 22 hours
To measure the pharmacokinetic parameters of taking avanafil with amlodipine | before dosing and after dosing at the hours of 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36, 48
  AUCc-tau Cmax Cmin Tmax AUC0-t AUC0-inf t1/2 Kel
To determine the effects of amlodipine on blood pressure and pulse rate | -0.5, -0.33, -0.17, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10 and 22 hours

CONTACTS AND LOCATIONS:
Overall Officials: Shiyin Yee, PhD, Study Director — VIVUS LLC
Locations (1):
- Celerion, Tempe, Arizona, United States